CLINICAL TRIAL: NCT04764526
Title: Can Protein-enriched Ice Cream Increase Protein- and Energy Intake and at the Same Time Evoke Positive Emotions - a Feasibility Study Among Hospitalized Older Patients
Brief Title: Ice Cream Enriched With Protein and Positive Emotions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inge Tetens (Other)
Responsible Party: Sponsor-Investigator, Inge Tetens, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: M238
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-04

CONDITIONS: Protein Intake
Keywords: Protein-enrichment; Older hospitalized patients

STUDY DESIGN:
Intervention Model Description: The participant will be their own control and will be randomised to start with control followed by intervention or the opposite order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein-enriched ice cream (Experimental): Two protein-enriched ice cream daily (afternoon and evening) in two days in addition to the normal menu
  Interventions: Other: Protein-enriched ice cream
- Control (No Intervention): Standard menu in two days

INTERVENTIONS:
Other: Protein-enriched ice cream — Offering two protein-enriched ice creams
  Arms: Protein-enriched ice cream

SUMMARY:
The primary aim is to investigate if protein-enriched ice cream has the feasibility to increase intake of protein without substituting other foods in hospitalized older patients and secondary, if the protein-enriched ice cream has the feasibility to increases the energy intake and evokes positive emotions in older hospitalized patients

DETAILED DESCRIPTION:
Methods/Design:

This study is conducted as a four days non-blinded randomised cross-over feasibility study with 24 hospitalized older patients. The intervention is conducted at the hospital. The intervention is two days with two protein-enriched ice cream daily with the aim of increasing the intake of protein and energy. The patients are asked to answer a questionnaire concerning the emotions the protein enriched ice cream evoke.The patients will be randomised to receive the standard menu the first two days followed by two days with standard menu plus protein-enriched ice cream or in the opposite order. The randomisation will be done by using sealed envelopes.

Recruitment:

Only admitted patients will be a part of the trial. The ward staff will identify the patients there are eligible to the trial as close as possible to the day of admission. The ward staff will ask those patients who meet the inclusion criteria if they will participate in the trail. The patients receive oral and written information on the trial and those who agree to participate are asked to sign a statement of consent before participating. The patients can at any time withdraw their consent and leave the trial.

Sample size:

The sample size is estimated to 24 patients, who will be their own control.

Statistical analysis:

Non-parametric statistical tests, median and range will be performed due to the small sample size and skew distribution. The Wilcoxon signed rank test for paired data, and Fisher's exact test for categorical data. Evoked emotion are measured as the percentages of patients who choose a particular emotion term.

ELIGIBILITY:
Inclusion Criteria:

- older admitted hospital patients age 65 or older, capable & Danish speaking (able to read and understand the oral and written information and give written consent), able to eat, eat ice cream and expected to stay at the hospital least four days.

Exclusion Criteria:

* terminally ill, tube feed, need of special diets, any medical indication suggesting that they should not participate or are on a weight reduction scheme

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Protein intake (g, %) | four consecutive days while hospitalized
  The change in protein intake with and without protein-enriched ice cream.

SECONDARY OUTCOMES:
Energy intake (kJ, %) | four consecutive days while hospitalized
  The change in energy intake with and without protein-enriched ice cream.
Evoked emotions | one day while hospitalized (first time the patients is offered a protein-enriched ice cream)
  Check-all-that-apply (CATA) emotions word questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Inge Tetens, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No